CLINICAL TRIAL: NCT07023094
Title: Comparison of Analgesic Efficacy of Pericapsular Nerve Group (PENG) Block With Lateral Femoral Cutaneous Nerve Block (LFCB) Versus Lumbar and Sacral Erector Spinae Plane Blocks (L-ESPB and S-ESPB) in Pediatric Hip Surgery: A Randomized Controlled Trial
Brief Title: PENG With LFCB vs. ESP Blocks for Pediatric Hip Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6/2025
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Hip Disease; Hip Dysplasia; Hip Arthropathy
MeSH Terms: conditions — Hip Dislocation | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG + LFCB (Active Comparator): U-S guided PENG block - 0.4ml/kg 0.2% ropivacaine
  + U-S guided LFCB - 0.1ml/kg 0.2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% for PENG Block; Drug: Ropivacaine 0.2% for LFCB
- L-ESPB + S-ESPB (Active Comparator): U-S guided L-ESPB - 0.25ml/kg 0.2% ropivacaine
  + U-S guided S-ESPB - 0.25ml/kg 0.2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% for L-ESPB; Drug: Ropivacaine 0.2% for S-ESPB

INTERVENTIONS:
Drug: Ropivacaine 0.2% for PENG Block — U-S guided PENG (0.4 mL/kg) with 0.2% ropivacaine
  Arms: PENG + LFCB
Drug: Ropivacaine 0.2% for LFCB — LFCB (0.1 mL/kg) with 0.2% ropivacaine
  Arms: PENG + LFCB
Drug: Ropivacaine 0.2% for L-ESPB — Lumbar ESPB (0.25ml/kg) with 0.2% ropivacaine
  Arms: L-ESPB + S-ESPB
Drug: Ropivacaine 0.2% for S-ESPB — Sacral ESPB (0.25ml/kg) with 0.2% ropivacaine
  Arms: L-ESPB + S-ESPB

SUMMARY:
This randomized controlled trial (RCT) compares the analgesic effectiveness of two regional anesthesia techniques-Pericapsular Nerve Group (PENG) block combined with Lateral Femoral Cutaneous Nerve Block (LFCB) versus Lumbar and Sacral Erector Spinae Plane Blocks (L-ESPB and S-ESPB)-in pediatric patients undergoing hip surgery.

DETAILED DESCRIPTION:
Orthopedic hip procedures in pediatric patients, including osteotomies, arthroscopic interventions, and reconstructive surgeries, often result in significant postoperative pain. Effective analgesia is critical for reducing surgical stress, accelerating rehabilitation, and minimizing opioid use and associated side effects. Regional anesthesia techniques have gained attention for their opioid-sparing effects and enhanced recovery profiles.

This randomized controlled trial aims to compare the analgesic effectiveness of two regional anesthetic approaches:

- The pericapsular nerve group (PENG) block is combined with the lateral fetal cutaneous nerve block (LFCB), targeting hip joint innervation directly and providing comprehensive sensory coverage.

Lumbar and sacral erector spinae plane blocks (L-ESPB and S-ESPB) employ fascial plane techniques to deliver analgesia by diffusing local anesthetic around nerves innervating the hip region.

This trial aims to establish the optimal regional anesthesia technique and determine the clinical benefits of using dexamethasone and dexmedetomidine as adjuvants. The results will guide clinicians toward evidence-based analgesic protocols in pediatric orthopedic hip surgery, potentially reducing opioid-related complications and improving patient recovery outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged between 2 and 16 years.
* Scheduled for elective orthopedic hip surgery, including: Osteotomies and Hip reconstruction surgeries
* ASA (American Society of Anesthesiologists) physical status classification: I-III.
* Written informed consent obtained from the patient's legal guardian(s).

Exclusion Criteria:

* Known allergy or hypersensitivity to any of the study medications
* Presence of infection or inflammation at the intended injection site(s) of regional anesthesia.
* Coagulopathy or bleeding disorders (including patients on anticoagulant therapy) that contraindicate nerve blocks.
* Neurological disorders or peripheral neuropathies that could influence sensory or motor assessment of the lower limbs.
* Cognitive impairment or behavioral disorders significantly affecting pain assessment accuracy or cooperation.
* History of chronic opioid use or known substance abuse.
* Severe systemic disease or condition compromising patient safety or interfering with study protocol adherence.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Opioid Consumption | 48 hours after surgery
  Total opiate consumption after surgery

SECONDARY OUTCOMES:
Time to first rescue opioid analgesia | 48 hours after surgery
  Time after surgery when the patient needs opiate for the first time
Numerical Rating Scale [range 0:10] | 4 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 8 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 12 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 24 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Numerical Rating Scale [range 0:10] | 48 hours after surgery
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
NLR | 12 hours after surgery
  neutrophile to lymphocyte ratio
NLR | 24 hours after surgery
  neutrophile to lymphocyte ratio
NLR | 48 hours after surgery
  neutrophile to lymphocyte ratio
PLR | 12 hours after surgery
  platelet to lymphocyte ratio
PLR | 24 hours after surgery
  platelet to lymphocyte ratio
PLR | 48 hours after surgery
  platelet to lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Reysner, M.D. Ph.D., Principal Investigator — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes